CLINICAL TRIAL: NCT06677502
Title: The Usefulness of Cerebrolysin in Alleviating the Severity of Delirium in Critically Ill Patients
Brief Title: Cerebrolysin in Critically Ill Patients With Delirium
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Wojciech Dąbrowski, Prof. MD, PhD, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEREBDEL; DS352/2024 (Other Grant/Funding Number: Medical University of Lublin, Poland)
Record Dates: First submitted 2024-09-29; First posted 2024-11-06 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Cognitive Impairment
Keywords: delirium; critically ill; treatment; Cerebrolysin
MeSH Terms: conditions — Cognitive Dysfunction; Delirium; Critical Illness | interventions — cerebrolysin

STUDY DESIGN:
Intervention Model Description: Patients enrolled to the intervention group (CER group) receive Cerebrolysin for 7 consecutive days at a dose of 50mL daily administrated in 250 mL 0.9% NaCl. Patients enrolled the control group (K group) receive 250 mL 0.9% NaCl.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cerebrolysin arm. (Experimental): Patients in group CER received Cerebrolysin infusion at the dose of 50 mL solved in 0.9% NaCl for seven consecutive days, after delirium diagnose.
  Interventions: Drug: Cerebrolysin
- Control arm. (Placebo Comparator): Patients in group K (control) received 0.9% NaCl for seven consecutive days.
  Interventions: Other: Saline Solution - IV

INTERVENTIONS:
Drug: Cerebrolysin — Patients were randomized into two groups: CBL - patients treated with cerebrolysin at the daily dose of 50 mL, and K - control patients treated without cerebrolysin. Cerebrolysin was administrated intravenously on the day the delirium was detected and then for seven consecutive days.
  Arms: Cerebrolysin arm.
Other: Saline Solution - IV — Patients enrolled in group K received the infusion of 0.9% Saline solution at a volume of 250 mL.
  Arms: Control arm.

SUMMARY:
Delirium is a severe problem in critically ill patients, and it is associated with increased morbidity, mortality, and extended stay in hospital. The pathophysiology of delirium is multifactorial and still poorly recognized. Several authors proposed different pathomechanisms of delirium. The most likely of these are a metabolic response to cerebral hypoxia/hyperoxia, oxidative stress with excessive reactive oxygen species production, neuroinflammation following general inflammatory response, disorders in neurotransmitters, especially impaired cholinergic and dopaminergic transmissions and dysregulation of tryptophan metabolisms including kynurenine and serotonin/melatonin pathways. The multifactorial pathomechanism of delirium significantly reduces targeted therapy. Due to cerebrolysin properties, it seems reasonable to conclude that this substance is effective in the prevention and treatment of delirium in critically ill patients. Cerebrolysin is commonly used in neurologic patients treated for dementia and Alzheimer's disease. It possesses antioxidative properties, which reduce the severity of post-ischaemic neuronal dysfunction and improve neuronal plasticity. It also increases acetylcholinesterase and butyrylcholinesterase in a dose-dependent manner, improving neuronal plasticity.

Additionally, cerebrolysin reduces neuroinflammation and neuronal cell apoptosis by activating toll-like receptor pathways. These properties closely correspond to the pathomechanism of delirium.

Therefore, the aim of this study is to analyze the effectiveness of treatment with Cerebrolysin in critically ill patients with delirium.

This study enrolls adult critically ill patients. Prior to delirium detection, the Richmond Agitation-Sedation Scale (RASS) is used to assess the level of consciousness. Patients with RASS-4 or -5 were excluded from the analysis, as these disorders of consciousness preclude the determination of the degree of delirium, which is a requisite component of the study. Delirium is detected by the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) and the Intensive Care Delirium Screening Checklist (ICDSC). Additionally, the Montreal Cognitive Assessment Scale is used to detect mild cognitive impairment. The primary endpoint of this study is an analysis of the prevalence and severity of delirium symptoms. The secondary endpoint is an analysis of the duration of delirium.

DETAILED DESCRIPTION:
This is an observational, interventional study. Adult critically ill patients treated with mechanical ventilation due to acute respiratory insufficiency complicating sepsis, septic shock, pneumonia, acute respiratory distress syndrome (ARDS) and polytrauma patients without traumatic brain injury are enrolled to this study. All patients should be treated in accordance with the most up-to date recommendations for the specific disease. None of the patients should be treated with neuroprotective medication before the diagnosis of delirium. Patients are randomized into two groups: CBL - patients treated with cerebrolysin and K - control patients treated without cerebrolysin. Cerebrolysin is administered in a daily dose of 50ml, dissolved in 0.9% NaCl. This mixture is infused for one hour. The treatment is initiated when the delirium is detected and continued for seven consecutive days.

The diagnosis of delirium is based on four principal criteria of the CAM-ICU test: 1/ Sudden onset of disturbance, 2/ Lack of focus of attention, 3/ Altered state of consciousness, and 4/ Disorganised thinking. Of these, criterion feature 2 is regarded as the most crucial in establishing a diagnosis of delirium.

The ICDSC method takes into account eight criteria which include: The ICDSC method considers eight criteria that include: 1/ any disturbance of consciousness (RASS other than 0), 2/ attention deficit disorder, 3/ disorientation, 4/ hallucinations, 5/ psychomotor agitation or retardation, 6/ speech or mood disturbances, 7/ disturbance of sleep-wake cycle, 8/ diurnal variability of symptoms. One point is added for each criterion. A score of 4 points or higher indicates a diagnosis of full-blown delirium, while a score of 1 to 3 points indicates subclinical delirium.

The initial detection of delirium using the CAM-ICU and ICDSC scales is conducted one to three days after the cessation of sedative infusion when the patient's sedation level reaches 3 on the RASS scale. Subsequent follow-up analysis is performed on days 7-8 after the diagnosis of delirium.

The MoCA test is performed in the days 7-8. The MoCA test is assessed using the Geriatric Assessment Tool Kit (https://geriatrictoolkit.missouri.edu) with the following points: 1/ Short term memory, 2/ Visuospatial abilities, 3/ Executive functions, 4/ attention and concentration, 5/ working memory, 6/ language, 7/ Orientation to time and place. A score of 24 points or less is the cut-off for mild cognitive impairment, while 19 points or less for dementia diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* age > 18,
* symptoms of delirium,
* critical illness treated in Intensive Care Unit

Exclusion Criteria:

* pregnancy
* traumatic brain injury,
* neuroinflammatory diseases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
CAM-ICU test | seven days
  Cerebrolysin, 50 mL daily administered intravenously for seven consecutive days, reduces or alleviates the severity of delirium detected by the CAM-ICU test.
ICDSC test | seven days
  Cerebrolysin, 50 mL daily administered intravenously for seven consecutive days, reduces or alleviates the severity of delirium detected by the ICDSC test.

SECONDARY OUTCOMES:
MoCA test | seven days
  Cerebrolysin infusion at the dose of 50 mL daily administrated intravenously reduces or alleviates the severity of cognitive impairment detected by the MoCA test.

CONTACTS AND LOCATIONS:
Locations (1):
- First Department of Anaesthesiology and Intensive Therapy Medical University of Lublin, Lubin, Lublin Voivodeship, Poland

REFERENCES:
- [Result] Nakanishi N, Liu K, Kawauchi A, Okamura M, Tanaka K, Katayama S, Mitani Y, Ota K, Taito S, Fudeyasu K, Masuka Y, Yoshihiro S, Utsumi S, Nishikimi M, Masuda M, Iida Y, Kawai Y, Hatakeyama J, Hifumi T, Unoki T, Kawakami D, Obata K, Katsukawa H, Sumita H, Morisawa T, Takahashi M, Tsuboi N, Kozu R, Takaki S, Haruna J, Fujinami Y, Nosaka N, Miyamoto K, Nakamura K, Kondo Y, Inoue S, Nishida O. Instruments to assess post-intensive care syndrome assessment: a scoping review and modified Delphi method study. Crit Care. 2023 Nov 7;27(1):430. doi: 10.1186/s13054-023-04681-6. PMID 37936249
- [Result] Smith HA, Gangopadhyay M, Goben CM, Jacobowski NL, Chestnut MH, Savage S, Rutherford MT, Denton D, Thompson JL, Chandrasekhar R, Acton M, Newman J, Noori HP, Terrell MK, Williams SR, Griffith K, Cooper TJ, Ely EW, Fuchs DC, Pandharipande PP. The Preschool Confusion Assessment Method for the ICU: Valid and Reliable Delirium Monitoring for Critically Ill Infants and Children. Crit Care Med. 2016 Mar;44(3):592-600. doi: 10.1097/CCM.0000000000001428. PMID 26565631
- [Result] Landoure G, Sullivan JM, Johnson JO, Munns CH, Shi Y, Diallo O, Gibbs JR, Gaudet R, Ludlow CL, Fischbeck KH, Traynor BJ, Burnett BG, Sumner CJ. Exome sequencing identifies a novel TRPV4 mutation in a CMT2C family. Neurology. 2012 Jul 10;79(2):192-4. doi: 10.1212/WNL.0b013e31825f04b2. Epub 2012 Jun 6. No abstract available. PMID 22675077
- [Result] Flores IO, Trevino S, Diaz A. Neurotrophic fragments as therapeutic alternatives to ameliorate brain aging. Neural Regen Res. 2023 Jan;18(1):51-56. doi: 10.4103/1673-5374.331867. PMID 35799508
- [Result] Hoel H, Heggelund L, Reikvam DH, Stiksrud B, Ueland T, Michelsen AE, Otterdal K, Muller KE, Lind A, Muller F, Dudman S, Aukrust P, Dyrhol-Riise AM, Holter JC, Troseid M. Elevated markers of gut leakage and inflammasome activation in COVID-19 patients with cardiac involvement. J Intern Med. 2021 Apr;289(4):523-531. doi: 10.1111/joim.13178. Epub 2020 Oct 8. PMID 32976665
- [Result] Sharma S, Raj K, Singh S. Protective effects of cerebrolysin against chemotherapy (carmustine) induced cognitive impairment in Albino mice. Drug Chem Toxicol. 2022 Nov;45(6):2769-2779. doi: 10.1080/01480545.2021.1991195. Epub 2021 Oct 21. PMID 34674598
- [Result] Liu Z, Hu M, Lu P, Wang H, Qi Q, Xu J, Xiao Y, Fan M, Jia Y, Zhang D. Cerebrolysin alleviates cognitive deficits induced by chronic cerebral hypoperfusion by increasing the levels of plasticity-related proteins and decreasing the levels of apoptosis-related proteins in the rat hippocampus. Neurosci Lett. 2017 Jun 9;651:72-78. doi: 10.1016/j.neulet.2017.04.022. Epub 2017 Apr 27. PMID 28458021
- [Result] Kotfis K, Ely EW, Shehabi Y. Intensive care unit delirium-a decade of learning. Lancet Respir Med. 2023 Jul;11(7):584-586. doi: 10.1016/S2213-2600(23)00222-9. No abstract available. PMID 37414511
- [Result] Ottens TH, Hermes C, Page V, Oldham M, Arora R, Bienvenu OJ 3rd, van den Boogaard M, Caplan G, Devlin JW, Friedrich ME, van Gool WA, Hanison J, Hansen HC, Inouye SK, Kamholz B, Kotfis K, Maas MB, MacLullich AMJ, Marcantonio ER, Morandi A, van Munster BC, Muller-Werdan U, Negro A, Neufeld KJ, Nydahl P, Oh ES, Pandharipande P, Radtke FM, Raedt S, Rosenthal LJ, Sanders R, Spies CD, Vardy ERLC, Wijdicks EF, Slooter AJC. The Delphi Delirium Management Algorithms. A practical tool for clinicians, the result of a modified Delphi expert consensus approach. Delirium (Bielef). 2024;2024:10.56392/001c.90652. doi: 10.56392/001c.90652. Epub 2024 Jan 12. PMID 38348284
- [Result] Kotfis K, Maj P, Szylinska A, Pankowiak M, Reszka E, Ely EW, Marra A. The spectrum of psychological disorders in family members of patients suffering from delirium associated with critical illness: a prospective, observational study. Sci Rep. 2024 Feb 24;14(1):4562. doi: 10.1038/s41598-024-53968-3. PMID 38402273
- [Result] Dabrowski W, Siwicka-Gieroba D, Gasinska-Blotniak M, Zaid S, Jezierska M, Pakulski C, Williams Roberson S, Wesley Ely E, Kotfis K. Pathomechanisms of Non-Traumatic Acute Brain Injury in Critically Ill Patients. Medicina (Kaunas). 2020 Sep 13;56(9):469. doi: 10.3390/medicina56090469. PMID 32933176
- [Result] Cui S, Chen N, Yang M, Guo J, Zhou M, Zhu C, He L. Cerebrolysin for vascular dementia. Cochrane Database Syst Rev. 2019 Nov 11;2019(11):CD008900. doi: 10.1002/14651858.CD008900.pub3. PMID 31710397
- [Result] Seidl LF, Aigner L. Comparing the biological activity and composition of Cerebrolysin with other peptide preparations. J Med Life. 2024 Jan;17(1):24-27. doi: 10.25122/jml-2024-0129. PMID 38737662
- [Result] Ulderich Williams SC, Qaddoumi AI, Meghreblian JT, McBride ME, King SA, Elahi MA, Tuggle D, Heidel RE, Smith LM. Incidence and Risk Factors for ICU-Associated Delirium in the Alert Geriatric Trauma Population. Am Surg. 2024 Jul;90(7):1866-1871. doi: 10.1177/00031348241241707. Epub 2024 Mar 23. PMID 38520278
- [Result] Duprey MS, Devlin JW, van der Hoeven JG, Pickkers P, Briesacher BA, Saczynski JS, Griffith JL, van den Boogaard M. Association Between Incident Delirium Treatment With Haloperidol and Mortality in Critically Ill Adults. Crit Care Med. 2021 Aug 1;49(8):1303-1311. doi: 10.1097/CCM.0000000000004976. PMID 33861548
- [Result] Lu W, Zhu Z, Shi D, Li X, Luo J, Liao X. Cerebrolysin alleviates early brain injury after traumatic brain injury by inhibiting neuroinflammation and apoptosis via TLR signaling pathway. Acta Cir Bras. 2022 Sep 5;37(6):e370605. doi: 10.1590/acb370605. eCollection 2022. PMID 36074398
- [Result] Kotfis K, Marra A, Ely EW. ICU delirium - a diagnostic and therapeutic challenge in the intensive care unit. Anaesthesiol Intensive Ther. 2018;50(2):160-167. doi: 10.5603/AIT.a2018.0011. Epub 2018 Jun 8. PMID 29882581
- [Result] Eman G, Marsh A, Gong MN, Hope AA. Utility of Screening for Cognitive Impairment at Hospital Discharge in Adult Survivors of Critical Illness. Am J Crit Care. 2022 Jul 1;31(4):306-314. doi: 10.4037/ajcc2022447. PMID 35773197